CLINICAL TRIAL: NCT01165684
Title: A Randomised, Controlled, Open Label, Multicentre, Multinational, Treat-to-target Trial Investigating the Efficacy and Safety of Intensification With Addition of Bolus Insulin Aspart in Subjects With Type 2 Diabetes Inadequately Controlled on Basal Insulin With or Without Oral Anti-diabetic Drugs: Step-wise Addition Versus Complete Basal-bolus Therapy
Brief Title: Efficacy and Safety of Basal-bolus Therapy, Comparing Stepwise Addition of Insulin Aspart Versus Complete Basal-bolus Regimen
Acronym: Full STEP™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-3786; 2010-018974-19 (EudraCT Number); U1111-1116-0908 (Other: WHO)
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Results first posted 2013-06-11 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Step-wise (Experimental)
  Interventions: Drug: insulin aspart; Drug: insulin detemir
- Basal-bolus (Active Comparator)
  Interventions: Drug: insulin aspart; Drug: insulin detemir

INTERVENTIONS:
Drug: insulin aspart — Insulin aspart added stepwise according to the largest meal following an evaluation of HbA1c.
  Doses individually adjusted.
  Arms: Step-wise
Drug: insulin aspart — Insulin aspart added before each main meal. Doses individually adjusted.
  Arms: Basal-bolus
Drug: insulin detemir — Insulin detemir as basal insulin, adminstered once daily. Doses individually adjusted.

SUMMARY:
This trial is conducted in Europe, and North and South America. The aim of this clinical trial is to investigate if the two treatments are equally effective.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for at least 12 months
* Basal insulin treatment (NPH once or twice daily, insulin glargine once daily or insulin detemir once daily) for at least 6 months
* HbA1c: 7.0-9.0 % (both inclusive) by central laboratory analysis (one retest analysed at the central laboratory within a week is permitted with the result of the last sample being conclusive)
* BMI (Body Mass Index) less than 40.0 kg/m^2

Exclusion Criteria:

* Previous use of pre-mix or bolus insulin (allowed is previous use of bolus insulin only in case of a hospitalisation or a severe condition requiring intermittent use of bolus insulin for less than 14 consecutive days, but not during the last 6 months prior to screening visit (Visit 1)
* Use of GLP-1 (Glucagon-like peptide-1) receptor agonists or pramlintide within the last 6 months prior to prior to screening visit (Visit 1)
* Anticipated change in concomitant medication known to interfere significantly with glucose metabolism (e.g. systemic corticosteroids, beta-blockers, MAO (Monoamine oxidase) inhibitors, etc.)
* Cardiovascular disease, within the last 12 months prior to screening visit (Visit 1), defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure sitting at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg). For Argentina: systolic blood pressure sitting at least 150 mmHg and/or diastolic blood pressure at least 90 mmHg
* Impaired liver function, defined as ALAT (Alanine aminotransferase) at least 2.5 times upper limit of normal (one retest analysed at the central laboratory within a week is permitted with the result of the last sample being conclusive)
* Impaired renal function defined as serum creatinine above 135 micromol/L (above 1.5 mg/dL) for males and above 110 micromol/L (above 1.2 mg/dL) for females; and, if required by the locally applicable metformin label, glomerular filtration rate below 60 ml/min, calculated by the Cockroft & Gault formula). One retest within a week is permitted with the result of the last sample being conclusive
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic episode, during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Proliferative retinopathy or maculopathy requiring treatment according to the Investigator
* Treatment with OADs (Oral anti-diabetic drug) contraindicated or unapproved for combination treatment with insulin (according to local OAD label)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (61):
- United States (31):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Scottsdale, Arizona
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Springfield, Massachusetts
  - Novo Nordisk Investigational Site, Brooklyn Center, Minnesota
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, Beavercreek, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Newport News, Virginia
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mendoza
- Brazil (5):
  - Novo Nordisk Investigational Site, Goiânia, Goiás
  - Novo Nordisk Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Campinas
  - Novo Nordisk Investigational Site, Porto Alegre
- Canada (11):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Coquitlam, British Columbia
  - Novo Nordisk Investigational Site, Langley, British Columbia
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Victoria, British Columbia
  - Novo Nordisk Investigational Site, Chatham, Ontario
  - Novo Nordisk Investigational Site, Kingston, Ontario
  - Novo Nordisk Investigational Site, Gatineau, Quebec
  - Novo Nordisk Investigational Site, Lachine, Quebec
  - Novo Nordisk Investigational Site, Mirabel, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
- France (5):
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Sète
  - Novo Nordisk Investigational Site, Vénissieux
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Slovenia (4):
  - Novo Nordisk Investigational Site, Brežice
  - Novo Nordisk Investigational Site, Kranj
  - Novo Nordisk Investigational Site, Novo Mesto
  - Novo Nordisk Investigational Site, Trbovlje

REFERENCES:
- [Result] Rodbard HW, Visco VE, Andersen H, Hiort LC, Shu DH. Treatment intensification with stepwise addition of prandial insulin aspart boluses compared with full basal-bolus therapy (FullSTEP Study): a randomised, treat-to-target clinical trial. Lancet Diabetes Endocrinol. 2014 Jan;2(1):30-7. doi: 10.1016/S2213-8587(13)70090-1. Epub 2013 Sep 25. PMID 24622667
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 69 sites in 7 countries: Argentina (7), Brazil (5), Canada (12), France (7), Macedonia (1), Slovenia (4), and the US (31). Of 12 sites in Canada, one site (Site 303) closed early on 07-Mar-2011.
Pre-assignment Details: Subjects on pre-trial metformin and pioglitazone continued their medication.
Groups:
- Step-wise: In addition to insulin detemir once daily, insulin aspart was added step-wise starting at the randomisation visit (Week 0) with the first bolus before the largest meal, followed by a second bolus at the second largest meal at Week 11 in subjects with HbA1c ≥ 7.0% at Week 10, and a second or third bolus at Week 22 in subjects with HbA1c ≥ 7.0% at Week 21. Subjects on pre-trial metformin and pioglitazone continued their medication.
- Basal-bolus: In addition to insulin detemir once daily, insulin aspart was added before each of the main meals (breakfast, lunch and dinner) starting at the randomisation visit. Subjects on pre-trial metformin and pioglitazone continued their medication.
Period: Overall Study
Arm/Group | Step-wise | Basal-bolus
Started | 201 | 200
Exposed | 198 (3 subjects withdrew prior to exposure to trial drug) | 199 (1 subject withdrew prior to exposure to trial drug)
Completed | 173 | 148
Not Completed | 28 | 52
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Protocol Violation | 7 | 15
Not completed — Withdrawal Criteria | 2 | 13
Not completed — Unclassified | 16 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Step-wise | Basal-bolus | Total
Number analyzed (Participants) | 201 | 200 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.1) | 59.6 (9.5) | 59.8 (9.3)
Gender [Count of Participants; unit: Participants]
  Female | 97 | 101 | 198
  Male | 104 | 99 | 203
Body weight [Mean (Standard Deviation); unit: kg] | 88.9 (18.7) | 86.1 (15.2) | 87.5 (17.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (4.8) | 30.7 (4.6) | 31.1 (4.7)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.9 (0.6) | 7.9 (0.6) | 7.9 (0.6)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 7.0 (1.9) | 6.9 (1.6) | 6.9 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline to Week 32
Description: Estimated mean change from baseline in HbA1c after 32 Weeks of treatment
Time Frame: Week 0, Week 32
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 383 subjects contributed to the statistical analysis at Week 32.
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 195 | 188
percentage of glycosylated haemoglobin | -0.98 (0.06) | -1.12 (0.06)
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% CI was below or equal to 0.4% or equivalently if the p-value for the one-sided test of was less than or equal to 2.5%, where D is the mean treatment difference (step-wise regimen minus basal-bolus regimen); p = 0.088, Regression, Linear; Estimated treatment difference, Mean = 0.14, 95% CI [-0.02 to 0.30]

2. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline to Week 10
Description: Estimated mean change from baseline in HbA1c after 10 Weeks of treatment
Time Frame: Week 0, Week 10
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 376 subjects contributed to the statistical analysis at Week 10.
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 193 | 183
percentage of glycosylated haemoglobin | -0.45 (0.05) | -1.00 (0.05)
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p < 0.001, Regression, Linear; Estimated treatment difference, Mean = 0.55, 95% CI [0.42 to 0.69]

3. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline to Week 21
Description: Estimated mean change from baseline in HbA1c after 21 Weeks of treatment
Time Frame: Week 0, Week 21
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 383 subjects contributed to the statistical analysis at Week 21.
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 195 | 188
percentage of glycosylated haemoglobin | -0.78 (0.06) | -1.15 (0.06)
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p < 0.001, Regression, Linear; Estimated treatment difference, Mean = 0.37, 95% CI [0.21 to 0.53]

4. Secondary Outcome: Proportion of Subjects Reaching Glycosylated Haemoglobin (HbA1c) Below 7.0% at Week 10
Description: Proportion of subjects reaching HbA1c below 7.0% at Week 10
Time Frame: Week 10
Population: as for outcome 2
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 193 | 183
percentage (%) of subjects | 19.2 | 56.3
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.85, 95% CI [4.12 to 11.39]

5. Secondary Outcome: Proportion of Subjects Reaching Glycosylated Haemoglobin (HbA1c) Below 7.0% at Week 21
Description: Proportion of subjects reaching HbA1c below 7.0% at Week 21
Time Frame: Week 21
Population: as for outcome 3
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 195 | 188
percentage (%) of subjects | 45.1 | 65.4
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.38, 95% CI [1.56 to 3.64]

6. Secondary Outcome: Proportion of Subjects Reaching Glycosylated Haemoglobin (HbA1c) Below 7.0% at Week 32
Description: Proportion of subjects reaching HbA1c below 7.0% at Week 32
Time Frame: Week 32
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 195 | 188
percentage (%) of subjects | 55.9 | 63.3
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p = 0.146, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI [0.90 to 2.07]

7. Secondary Outcome: Fasting Plasma Glucose (FPG) at Week 10
Description: Mean FPG at Week 10
Time Frame: Week 10
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 368 subjects contributed to data at Week 10.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 186 | 182
mmol/L | 7.1 (1.9) | 6.7 (1.9)

8. Secondary Outcome: Fasting Plasma Glucose (FPG) at Week 21
Description: Mean FPG at Week 21
Time Frame: Week 21
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 383 subjects contributed to the data at Week 21.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 195 | 188
mmol/L | 7.1 (2.3) | 7.0 (2.3)

9. Secondary Outcome: Fasting Plasma Glucose (FPG) at Week 32
Description: Estimated Mean FPG at Week 32
Time Frame: Week 32
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 195 | 188
mmol/L | 7.12 (0.17) | 7.01 (0.17)
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p = 0.635, Regression, Linear; Estimated Mean = 0.12, 95% CI [-0.37 to 0.60]

10. Secondary Outcome: Mean Plasma Glucose Increment Over 3 Meals (Breakfast, Lunch and Dinner) at Week 10
Description: Mean plasma glucose increment over 3 meals (breakfast, lunch and dinner) at Week 10
Time Frame: Week 10
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 326 subjects contributed to the data at Week 10.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 165 | 161
mmol/L | 2.3 (2.2) | 1.4 (2.0)

11. Secondary Outcome: Mean Plasma Glucose Increment Over 3 Meals (Breakfast, Lunch and Dinner) at Week 21
Description: Mean plasma glucose increment over 3 meals (breakfast, lunch and dinner) at Week 21
Time Frame: Week 21
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 343 subjects contributed to the data at Week 21.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 176 | 167
mmol/L | 1.9 (1.8) | 1.5 (1.8)

12. Secondary Outcome: Mean Plasma Glucose Increment Over 3 Meals (Breakfast, Lunch and Dinner) at Week 32
Description: Estimated mean plasma glucose increment over 3 meals (breakfast, lunch and dinner) at Week 32
Time Frame: Week 32
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 352 subjects contributed to the statistical analysis at Week 32.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 182 | 170
mmol/L | 1.64 (0.12) | 1.28 (0.13)
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p = 0.046, Regression, Linear; Estimated mean = 0.36, 95% CI [0.01 to 0.71]

13. Secondary Outcome: Body Weight at Week 32
Description: Estimated mean body weight after 32 Weeks of treatment
Time Frame: Week 32
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). 378 subjects contributed to the statistical analysis at Week 32.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 190 | 188
kg | 89.32 (0.28) | 89.80 (0.28)
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p = 0.228, Regression, Linear; Estimated mean = -0.48, 95% CI [-1.25 to 0.30]

14. Secondary Outcome: Body Mass Index (BMI) at Week 32
Description: Estimated mean BMI after 32 Weeks of treatment
Time Frame: Week 32
Population: as for outcome 13
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 190 | 188
kg/m^2 | 31.86 (0.10) | 32.03 (0.10)
Statistical Analysis 1: Comparison: Step-wise vs Basal-bolus; Test type: Superiority or Other; p = 0.224, Regression, Linear; Estimated mean = -0.17, 95% CI [-0.45 to 0.11]

15. Secondary Outcome: Hypoglycaemic Episodes (Rate of All Treatment Emergent Hypoglycaemia Episodes)
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of exposure to randomised treatment and no later than 1 day after the last day of randomised treatment.
Time Frame: Week 0 to Week 32
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator. 397 subjects contributed with data.
Measure: Number; unit: Episodes /year of patient exposure
Arm/Group | Step-wise | Basal-bolus
Number analyzed (Participants) | 198 | 199
Episodes /year of patient exposure | 33.47 | 57.56

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time of consent until 32 weeks of treatment and if needed were followed up after the final visit
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator
Arm/Group | Step-wise | Basal-bolus
Serious Adverse Events (participants affected / at risk) | 18/198 | 15/199
Other Adverse Events (participants affected / at risk) | 40/198 | 47/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Step-wise (N=198) | Basal-bolus (N=199)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial translocation (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 5 (6)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 3 (3)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Step-wise (N=198) | Basal-bolus (N=199)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 10 (10)
Oedema peripheral (General disorders) | 4 (5) | 10 (10)
Influenza (Infections and infestations) | 10 (11) | 13 (14)
Nasopharyngitis (Infections and infestations) | 16 (19) | 13 (18)
Headache (Nervous system disorders) | 10 (15) | 11 (13)

LIMITATIONS AND CAVEATS:
A higher proportion of subjects did not complete the trial in the basal-bolus arm (52 subjects, 26.0%) than in the step-wise arm (28 subjects, 13.9%).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Novo Nordisk reserves the right to prior review of such publications and to ask for delay of publication of individual site results until after the primary manuscript is accepted for publication.